CLINICAL TRIAL: NCT06412146
Title: Diabetes Link Discord
Brief Title: Children's Mercy Teens With Type 1 Diabetes Will Participate in an Online Peer Support Group.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00003114
Record Dates: First submitted 2024-04-18; First posted 2024-05-14 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Support Group (Experimental)
  Interventions: Behavioral: Peer Support Group

INTERVENTIONS:
Behavioral: Peer Support Group — Participation in an Online Peer Support Group

SUMMARY:
The goal of this observational study is to examine the impact of an online peer support group in Children's Mercy teens with Type 1 Diabetes.

The main objectives are to examine the feasibility and acceptability of the Diabetes Link's online social platform Discord among youth with diabetes as it relates to peer support, diabetes management, and usability and to examine the efficacy/magnitude of the effect of the Discord group on treatment adherence among youth with diabetes.

Participants will participate in an online peer support group for 3 months and provide their feedback while doing so.

ELIGIBILITY:
Inclusion Criteria:

* T1D Diagnosis
* 16-19 years old
* 11th-12th graders
* Access to smartphone/laptop
* English-speaking

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Support Group
Started | 10
Completed | 6
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Though 10 consented to the study, only 4 individuals participated in the group events and posts, and only 5 individuals completed the final survey.
Arm/Group | Peer Support Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Discord User Metrics
Description: Participant involvement was measured by the number of user instances of involvement in the online group (group chats plus online events attended).
Time Frame: 3 months
Population: Of the 10 who consented to the study, only 4 participated in chats and online events.
Measure: Median (Inter-Quartile Range); unit: instances
Arm/Group | Peer Support Group
Number analyzed (Participants) | 4
instances | 12.5 [8.5 to 45]

2. Primary Outcome: "Yes" Responses on Final Feedback Survey
Description: Each participant had 4 yes/no questions to answer about their study experience. "Yes" implied high satisfaction, and "no" meant there was room for improvement.
Time Frame: 3 months
Population: Of the 10 participants who consented to the study, only 4 completed the final survey.
Measure: Median (Inter-Quartile Range); unit: responses
Arm/Group | Peer Support Group
Number analyzed (Participants) | 4
responses | 3.5 [2.5 to 4]

3. Secondary Outcome: Diabetes Measures
Description: percentage of HbA1c
Time Frame: 3 months
Population: Of the 4 participants who actively made posts and attended events in the online group, there was one participant for whom the HbA1c before and after gap is larger than the 180 days typically used in intervention analyses, and the dates of the before and after A1c measurements do not align with the intervention timing. So the HbA1c was examined for the other 3 participants.
Measure: Mean (Full Range); unit: percentage of HbA1c
Arm/Group | Peer Support Group
Number analyzed (Participants) | 3
percentage of HbA1c | 7.167 [6.6 to 7.6]

ADVERSE EVENTS:
Time Frame: approximately 3 months
Description: This was a minimal risk study.
Arm/Group | Peer Support Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT06412146/Prot_000.pdf